CLINICAL TRIAL: NCT01261156
Title: An Open-label, Single-Sequence Study to Evaluate the Effects of Diltiazem, a Moderate CYP3A4/A5 Inhibitor, on the Pharmacokinetics and Pharmacodynamics of E5555 and Its Metabolites in Healthy Subjects
Brief Title: A Study to Evaluate the Effects of Diltiazem, a Moderate CYP3A4/A5 Inhibitor, on the Pharmacokinetics and Pharmacodynamics of E5555 and Its Metabolites in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: E5555-A001-022
Record Dates: First submitted 2010-11-16; First posted 2010-12-16 (Estimated); Last update posted 2014-07-11 (Estimated); Status verified 2014-07

CONDITIONS: Healthy Subjects
MeSH Terms: interventions — E 5555; Diltiazem

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Study Arm 1 (Experimental)
  Interventions: Drug: E5555 100 mg and diltiazem
- Study Arm 2 (Experimental)
  Interventions: Drug: E5555 300 mg and diltiazem

INTERVENTIONS:
Drug: E5555 100 mg and diltiazem — E5555 single 100 mg oral dose in Treatment Period 1 Day 1 and in Treatment Period 2 Day 8. Diltiazem 360 mg orally each day for 14 days (Days 1-14) in Treatment Period 2.
  Arms: Study Arm 1
Drug: E5555 300 mg and diltiazem — E5555 single 300 mg oral dose in Treatment Period 1 and in Treatment Period 2 Day 8. Diltiazem 360 mg orally each day for 14 days (Days 1-14) in Treatment Period 2.
  Arms: Study Arm 2

SUMMARY:
The purpose of this study is to evaluate the effects of diltiazem on the pharmacokinetics (PK) and pharmacodynamics (PD) of E5555 and its metabolites in healthy subjects.

DETAILED DESCRIPTION:
This is an open-label, 2-arm study to evaluate the effects of diltiazem given in conjunction with E5555 on the PK of diltiazem and its metabolites. This is a Phase 1 study of 24 healthy male and female subjects that will be conducted at a single site. The planned duration of treatment for each subject is approximately 15 days including 1 day in Treatment Period 1 and 14 days in Treatment Period 2.

ELIGIBILITY:
Inclusion:

* Provide written informed consent
* Healthy, non-smoking, male or female subjects aged greater than or equal to 18 years to 55 years
* Body mass index (BMI) greater than or equal to 18 and less than or equal to 32 kg/m2 at Screening
* All females must have a negative serum beta human chorionic gonadotropin test result at Screening and Baseline. Females of child-bearing potential must agree to use a medically acceptable method of contraception commencing at least one menstrual cycle prior to starting study drug, throughout the entire study period and for 90 days after study drug discontinuation. The only subjects who will be exempt from this requirement are postmenopausal women or subjects who have been surgically sterilized or who are otherwise proven sterile.
* Male subjects who are partners of women of childbearing potential and are not abstinent or have not undergone a successful vasectomy must use, or their partners must use, a highly effective method of contraception commencing at least one menstrual cycle prior to starting study drug, throughout the entire study period and for 90 days after study drug discontinuation.
* Are willing and able to comply with all aspects of the protocol.

Exclusion:

* A family history, past medical history or clinical signs or symptoms of a bleeding diathesis
* History of any medical condition which will result in an increased risk of bleeding including but not limited to active or recurrent gastric ulcers, recent head trauma or surgery, severe hypertension, bacterial endocarditis etc
* Subjects with a history of spontaneous gum bleeding or clinical signs or symptoms on physical exam
* Clinically significant ocular disease or untreated visual or ocular symptoms
* Clinically significant abnormal electrocardiograms ECGs prior to dosing (Screening or Baselines) including a QT interval corrected for heart rate using Fredericia's formula (QTcF) and/or Bazett's formula (QTcB) greater than 450 ms
* Any history or past medical condition that will result in QTc prolongation or tachyarrhythmia such as Torsades de Points (includes hypokalemia, known family history of long QT syndrome, or any other known risk factors for Torsades de Points)
* A platelet count less than 150,000 or greater than 390,000 per mL at Screening or Baseline Period 1
* Abnormal (less than 80%) arachidonic acid induced platelet aggregation at Baseline Period 1
* History of unexplained syncope, hepato-bliary disease, sinus bradycardia, heart blocks, sick-sinus syndrome, cardiogenic shock, heart failure, seizures, or chronic obstructive lung disease
* Subjects with hypotension (less than 90 mm Hg systolic) and bradycardia (HR less than 40 beats per minute) or symptomatic bradycardia (HR less than 50 beats per minute)
* Received blood, donated blood, or experienced significant blood loss within 60 days prior to check-in
* Hypersensitivity to diltiazem or related compounds or ingredients in the formulation

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2010-10; Primary Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Evaluate the effects of diltiazem on the pharmacokinetics (PK ie. Cmax, Tmax, AUC and half-life) of E5555 and its known metabolites. | 18 days
Evaluate the effects of diltiazem on the thrombin- and thrombin receptor activating peptide (TRAP) -induced platelet aggregation of E5555 and its known metabolites | 18 days

SECONDARY OUTCOMES:
To evaluate the effects of co-adminstration of diltiazem and E5555 on the PK(ie. Cmax, Tmax, AUC and half-life) of diltiazem and its metabolites | 18 days
To evaluate effects of co-adminstration of diltiazem and E5555 on QTcF compared to E5555 alone | 18 days
To assess safety and tolerability of a single dose of E5555 when given alone or in combination with diltiazem by recording the number of all adverse events following drug administration | 18 days

CONTACTS AND LOCATIONS:
Overall Officials: Chukwuemeka Okereke, Study Director — Eisai Limited
Locations (1):
- PRA International, Zuidlaren, Netherlands, Netherlands